CLINICAL TRIAL: NCT00395109
Title: PET/CT to Image Hypoxia in Head and Neck Tumours
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: R-06-370; 12660
Record Dates: First submitted 2006-11-01; First posted 2006-11-02 (Estimated); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Head and Neck Cancer
Keywords: cancer; hypoxia; PET scan; CT scan
MeSH Terms: conditions — Head and Neck Neoplasms; Neoplasms; Hypoxia | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: PET/CT — All study participates will be scanned with PET/CT scan before surgery.

SUMMARY:
Patients with head and neck cancer will be imaged with PET scan and CT scan in order to determine areas of the tumour that are hypoxic.

It is hypothesized that PET /CT will provide information on hypoxia of the tumors and tumor regions in head and neck cancer patients.

DETAILED DESCRIPTION:
Patients with head and neck cancer greater than 3 cm will imaged with PET scan and CT scan in order to determine areas of the tumour that are hypoxic. Following surgical removal, samples of the tumour will be evaluated for the expression of hypoxia genes. The preoperative imaging will be compared to the "gold standard" measures of hypoxic response at the level of gene transcription and a new hypoxia marker with the hypoxyprobe detection system (pimonidazole).

Hypothesis: FDG/PET visualization of glycolysis combined with CT visualization of blood flow will correlate with cellular response to hypoxic stress in head and neck tumors and intra-tumor regions. Measurement of relative levels of mRNAs encoding hypoxia response genes will be performed in cells microdissected from the surgical samples. Good correlation between imaging signals and direct molecular measures of hypoxic response in primary human tumors will provide information necessary to develop treatment strategies that employ targeted, increased radiation to hypoxic tumors.

Pimonidazole is an exogenous nitro-imidazole marker, which can be detected through immunohistochemical analysis of frozen sections. It detects cellular hypoxia upon becoming reduced in cells with low oxygen tension, a property that can be detected through antibody mediated detection of the reduced form. It has also shown to reliably and specifically stain hypoxic regions within the tumor, and to correlate well with patient prognosis and treatment outcome.

ELIGIBILITY:
Inclusion Criteria:

* All patients with head and neck tumours (>3cm diameter) without bone involvement.

Exclusion Criteria:

* Known allergy to contrast agents
* Poor kidney function (serum creatinine level > 2.0 mg/dL or 177 mmol/L)
* Pregnancy
* Breast-feeding
* Unable to lie supine
* Patient who were biopsied or operated upon within the past month.
* Patient who were treated with chemotherapy or radiation within the past month.
* Tumors that were obscured by artifacts (e.g. tooth fillings) in CT scans.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2006-11-08 (Actual); Primary Completion 2009-11-30 (Actual); Study Completion 2009-12-31 (Actual)

PRIMARY OUTCOMES:
FDG/PET visualization of glycolysis/blood flow in tumors and intra-tumor regions; | 2 years
Measurement of mRNAs levels encoding hypoxia response genes in tumor samples. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: John Yoo, MD, Principal Investigator — Dept. of Otolaryngology, London Health Science Center, London, Ontario, Canada
Locations (1):
- London Health Science Center, London, Ontario, Canada